CLINICAL TRIAL: NCT02639182
Title: A Multi-Center, Open Label, Randomized Phase 2 Study of AGS-16C3F vs. Axitinib in Metastatic Renal Cell Carcinoma
Brief Title: A Study of AGS-16C3F vs. Axitinib in Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGS-16C3F-15-3
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Axitinib; Metastatic Renal Cell Carcinoma; AGS-16C3F
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — AGS-16C3F; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGS-16C3F (Experimental): Participants received 1.8 milligram per kilogram (mg/kg) of AGS-16C3F once every three weeks by single intravenous (IV) infusion.
  Interventions: Drug: AGS-16C3F
- Axitinib (Active Comparator): Participants received 2 to 10 milligram (mg) of axitinib twice daily by oral administration as defined in the product label and per local institutional guidelines.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: AGS-16C3F — Intravenous (IV) infusion
  Arms: AGS-16C3F
Drug: Axitinib — Oral
  Other Names: Inlyta®
  Arms: Axitinib

SUMMARY:
The purpose of this study was to evaluate the progression free survival (PFS), based on investigator radiologic review, of AGS-16C3F compared to axitinib in subjects with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of RCC

  * Non-clear subjects must be ENPP3 positive, defined as IHC H-score ≥15
* Has evidence of progression on or after the last regimen received:

  * Clear cell subject: must have received at least 2 prior systemic regimens, one of which is an anti-VEGF agent.
  * Non-clear cell subject: must have received at least one prior anti-VEGF regimen
* Has measurable disease according to Response Criteria for Solid Tumors (RECIST v.1.1)
* Has Eastern Cooperative Group (ECOG) performance status of 0 or 1
* Has archive tumor tissue from primary tumor or metastatic site (excluding bone), for which the source and availability have been confirmed.

  * If no archive tissue is available, the subject may elect to have a biopsy performed to obtain tissue.
* Has adequate organ function including:

  * Hematopoietic function as follows:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L
    2. Platelet count ≥ 100 x 10 9/L
    3. Hemoglobin ≥ 9 g/dL (transfusions are allowed)
  * Renal Function as follows:

    1. Creatinine ≤ 1.5 x upper limit of normal (ULN), or calculated glomerular filtration rate (GFR) > 40 mL/min (Cockcroft-Gault) if creatinine > 1.5x ULN
  * Hepatic function, as follows:

    1. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5x ULN if known liver metastases
    2. Total bilirubin ≤ 1.5 x ULN
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) levels ≤1.5 x ULN. If institution does not report PT value, the international normalization ratio (INR) must be ≤ ULN.

  * If subject is receiving Coumadin (warfarin), a stable international normalization ratio (INR) of 2-3 is required.
* No clinical symptoms of hypothyroidism
* Urine Protein to Creatinine Ratio (uPCR) < 2.0

  * If uPCR ≥ 2.0 then a 24-hour urine collection can be performed to qualify. If this is performed to qualify, the protein result must be < 2 g per 24 hours.
* Female subject must either:

  * Be of non-childbearing potential:

    1. post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
    2. documented surgically sterile
  * Or, if of childbearing potential,

    1. Agree not to try to become pregnant during the study and for 6 months after the final study drug administration
    2. And have a negative serum pregnancy test ≤ 10 days of cycle 1, day 1 (C1D1)
  * And, if heterosexually active, agree to consistently use 2 forms of highly effective birth control* (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 6 months after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception* consisting of 2 forms of birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 6 months after the final study drug administration
* Male subject must not donate sperm starting at Screening and throughout the study period and, for 6 months after the final study drug administration

Note: *Highly effective forms of birth control include:

* Consistent and correct usage of established oral contraception.
* Established intrauterine device (IUD) or intrauterine system (IUS).
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

* Has previously been treated with axitinib, AGS-16C3F, or AGS-16M8F
* Has untreated brain metastasis. In the case of a solitary brain metastasis which has been resected, there must be evidence of a disease-free interval of at least 3 months post-surgery. For brain metastases treated with whole brain or stereotactic radiation therapy, brain imaging must be stable > 3 months. All subjects previously treated for brain metastases must be stable off corticosteroid therapy for at least 28 days prior to C1D1.
* Has uncontrolled hypertension defined as blood pressure > 150/90 on medication(s) by 2 blood pressure readings taken at least 1 hour apart.
* Has gastrointestinal abnormalities including:

  * inability to take oral medication;
  * requirement for intravenous alimentation;
  * prior surgical procedures affecting absorption including total gastric resection;
  * active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
  * malabsorption syndromes such as celiac disease, cystic fibrosis, inflammatory bowel disease, systemic sclerosis, and carcinoid syndrome
* Has ocular conditions such as:

  * Active infection or corneal ulcer
  * Monocularity
  * Visual acuity of 20/70 or worse in both eyes
  * History of corneal transplantation
  * Contact lens dependent (if using contact lens, must be able to switch to glasses during the entire study duration)
  * Uncontrolled glaucoma (topical medications allowed)
  * Uncontrolled or active ocular problems (e.g., retinopathy, macular edema, active uveitis, wet macular degeneration) requiring surgery, laser treatment, or intravitreal injections
  * Papilledema or other active optic nerve disorder
* Has used any investigational drug (including marketed drugs not approved for this indication) ≤ 14 days of C1D1. No time limit applies to the use of marketed drugs approved for this indication provided that the subject has progressed on the treatment and all toxicities attributable to the drug have resolved, returned to baseline or stabilized.
* Has known sensitivity to any of the ingredients of:

  * investigational product AGS-16C3F and/or,
  * Inlyta® (axitinib) and/or,
  * 1% prednisolone acetate ophthalmic suspension and any other corticosteroids.
* Is currently using (i.e., within 14-days prior to first dose) drugs that are known strong CYP3A4/5 inhibitors / inducers.
* Thromboembolic event (e.g., deep vein thrombosis [DVT] and pulmonary embolism [PE]) ≤ 4 weeks of C1D1.

  * Subjects who had a thromboembolic event ≤ 4 weeks of C1D1 must be receiving adequate anticoagulation treatment for at least 2 weeks before C1D1 and must continue as clinically indicated post first dose
* Has history bleeding disorders (e.g., pulmonary hemorrhage, significant hemoptysis, menometrorrhagia not responding to hormonal treatment) ≤ 2 months before C1D1
* Has active angina or Class III or IV Congestive Heart Failure (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 6 months of randomization, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, congestive heart failure, or arrhythmias not controlled by medication.
* Had major surgery ≤ 4 weeks of C1D1
* Is pregnant (confirmed by positive serum pregnancy test) or lactating
* Has active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) ≤ 10 days of C1D1
* Is unwilling or unable to comply with study requirements
* Has any medical or psychiatric disorder that compromises the ability of the subject to give written informed consent, and/or comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (26):
- United States (20):
  - Site US01026, Tucson, Arizona
  - Site US01008, La Jolla, California
  - Site US01007, Los Angeles, California
  - Site US01020, Los Angeles, California
  - Site US01019, Palo Alto, California
  - Site US01010, Atlanta, Georgia
  - Site US01023, Baltimore, Maryland
  - Site US01002, Boston, Massachusetts
  - Site US01004, Ann Arbor, Michigan
  - Site US01013, Detroit, Michigan
  - Site US01012, Omaha, Nebraska
  - Site US01006, Buffalo, New York
  - Site US01022, Durham, North Carolina
  - Site US01017, Portland, Oregon
  - Site US01021, Pittsburgh, Pennsylvania
  - Site US01011, Charleston, South Carolina
  - Site US01003, Houston, Texas
  - Site US01014, Temple, Texas
  - Site US01001, Seattle, Washington
  - Site US01009, Milwaukee, Wisconsin
- Canada (6):
  - Site CA02006, Calgary, Alberta
  - Site CA02004, Edmonton, Alberta
  - Site CA02005, Kelowna, British Columbia
  - Site CA02001, Vancouver, British Columbia
  - Site CA02002, Hamilton, Ontario
  - Site CA02008, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=AGS-16C3F-15-3
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14554&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were atleast 18 years of age with all histologies of confirmed renal cell carcinoma and evidence of progression on or after the last regimen received were enrolled.
Pre-assignment Details: Randomization was stratified by Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1), the number of prior systemic RCC regimens (2 or > 2) and Renal cell carcinoma (RCC), histology (clear or nonclear cell).
Groups:
- AGS-16C3F: Participants received 1.8 milligram per kilogram (mg/kg) of AGS-16C3F once every three weeks by single (60-minute) intravenous (IV) infusion.
- Axitinib: Participants received axitinib at a starting dose of 5 milligram (mg) orally twice daily and then adjusted to 2 to 10 mg orally twice daily, as defined in the product label and per local institutional guidelines.
Period: Overall Study
Arm/Group | AGS-16C3F | Axitinib
Started | 67 | 66
Treated | 66 | 65
Completed | 0 | 0
Not Completed | 67 | 66
Not completed — Disease Progression | 50 | 49
Not completed — Adverse Event | 7 | 5
Not completed — Physician Decision | 3 | 3
Not completed — Withdrew Consent | 5 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study Closure | 1 | 2
Not completed — Sponsor Ended Study | 0 | 1
Not completed — Randomized But Did Not Receive Study Drug | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who were randomized to study drug.
Groups:
- AGS-16C3F: Participants received 1.8 mg/kg of AGS-16C3F once every three weeks by single (60-minute) IV infusion.
- Axitinib: Participants received axitinib at a starting dose of 5 mg orally twice daily and then adjusted to 2 to 10 mg orally twice daily, as defined in the product label and per local institutional guidelines.
- Total: Total of all reporting groups
Arm/Group | AGS-16C3F | Axitinib | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (9.1) | 61.1 (8.9) | 61.7 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 49 | 49 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 64 | 62 | 126
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 59 | 56 | 115
  Race: Asian | 6 | 7 | 13
  Race: American Indian or Alaska Native | 1 | 1 | 2
  Race: Other | 1 | 2 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants were categorized based on ECOG Performance status 0 (Fully active, able to carry on all predisease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work))
  Participants
    0 | 19 | 19 | 38
    1 | 48 | 47 | 95
Histological Type [Count of Participants; unit: Participants]
  Clear cell | 55 | 55 | 110
  Non-clear cell | 12 | 11 | 23
Prognostic Risk Group [Count of Participants; unit: Participants] — Prognostic Risk Group reported based on Hengs's criteria.
  Participants
    Favorable (0 risk factors) | 5 | 10 | 15
    Intermediate (1-2 risk factors) | 48 | 43 | 91
    Poor (>=3 risk factors) | 14 | 13 | 27
Number of Prior Systemic Renal cell carcinoma (RCC) Treatment Regimens [Count of Participants; unit: Participants]
  2 if clear cell or 1 if non-clear cell histology | 35 | 33 | 68
  >2 if clear cell or >1 if non-clear cell histology | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Investigator Radiologic Review
Description: PFS was defined as the time from the date of randomization to the earliest of documented disease progression as defined by RECIST v.1.1 or death from any cause. PFS was analysed using Kaplan-Meier estimates. Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters (longest for non-nodal lesions, short axis for nodal lesions) of the target lesions taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of 1 or more new lesions is also considered progression. Participants were censored if there were 2 or more than 2 consecutive missing assesments immediately prior to death or progression; or no death and no postebaseline assesments; or if ininitiated non protocol anticancer treatment prior to death or prior to documentation of disease progression; or alive and not progressed.
Time Frame: From date of randomization to the earliest of either documented disease progression or death from any cause (up to 53 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Months | 2.9 [2.0 to 4.0] | 5.7 [5.3 to 9.1]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority — The difference between treatment groups was tested using a stratified log rank test at a one-sided 0.1 significance level; p = 0.983, Log Rank — The stratification factors were the ECOG PS at baseline and the number of prior systemic renal cell carcinoma (RCC) regimens, without any other covariate(s). The model contained terms for treatment group and stratum

2. Secondary Outcome: PFS Per RECIST v1.1 as Assessed by Blinded Central Radiology Assessment
Description: PFS was defined as the time from the date of randomization to the earliest of documented disease progression as defined by RECIST v.1.1 or death from any cause. PFS was analysed using Kaplan-Meier estimates. PD was defined as at least a 20% increase in the sum of diameters (longest for non-nodal lesions, short axis for nodal lesions) of the target lesions taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of 1 or more new lesions is also considered progression. Participants were censored if there were 2 or more than 2 consecutive missing assessments immediately prior to death or progression; or no death and no postebaseline assessments; or if initiated non protocol anticancer treatment prior to death or prior to documentation of disease progression; or alive and not progressed.
Time Frame: From date of randomization to the earliest of either documented disease progression or death from any cause (up to 40 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Months | 3.5 [2.1 to 3.8] | 4.5 [3.5 to 7.6]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.110, Log Rank — The stratification factors were the ECOG PS at baseline and the number of prior systemic RCC regimens, without any other covariate(s). The model contained terms for treatment group and stratum; Hazard Ratio (HR) = 1.423, 95% CI 2-sided [0.924 to 2.192]

3. Secondary Outcome: Objective Response Rate (ORR) Based on the Investigator's Radiographic Assessment
Description: ORR was defined as the percentage of participants who had a best overall response of complete response (CR) or partial response (PR). CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) with reduction in short axis to <10mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Time Frame: From date of randomization until data cutoff date of 21 August 2019 (up to 40 months)
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Percentage of Participants | 7.5 [2.5 to 16.6] | 18.2 [9.8 to 29.6]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority; p = 0.062, Cochran-Mantel-Haenszel — A Cochran-Mantel-Haenszel (CMH) analysis of the ORR, stratified for baseline ECOG-PS and number of prior systemic therapies for RCC, was conducted at a two-sided significance level of 0.05; Stratified Mantel-Haenszel estimate of the odds ratio for experiencing objective response, with the axitinib arm as the reference level, was reported; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.1 to 1.1]

4. Secondary Outcome: Duration of Response (DOR) Based on the Investigator's Radiographic Assessment
Description: DOR was defined as the time from the date of the first response of CR or PR (whichever was first recorded) to the first date of documented PD or death due to any cause. DOR was analysed using Kaplan-Meier estimates. CR and PR were defined in outcome measure 3 and PD was defined in outcome measures 1 and 2. Participants were censored if there were 2 or more than 2 consecutive missing assesments immediately prior to death or progression; or no death and no postebaseline assesments; or if ininitiated non protocol anticancer treatment prior to death or prior to documentation of disease progression; or alive and not progressed.
Time Frame: From date of first objective response until data cutoff date of 21 August 2019 (up to 40 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Months | 6.8 [3.8 to 18.4] | 6.7 [1.8 to 9.2]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority; p = 0.439, Log Rank — [p-value comment as in outcome 2, analysis 1]; The difference between treatment groups was tested using a stratified log rank test at a one-sided 0.1 significance level; Hazard Ratio (HR) = 0.376, 95% CI [0.031 to 4.482]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. OS was analysed using Kaplan-Meier estimates. Participants were censored if there was no death and no postbaseline contact or no death and at least one postbaseline follow-up.
Time Frame: Date of randomization until the date of death from any cause (up to 53 months)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Months | 13.1 [10.1 to 23.0] | 15.5 [12.7 to 21.6]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority; p = 0.746, Log Rank — Test conducted at a 2-sided significance level of 0.05. The stratification factors were the ECOG PS at baseline and number of prior systemic RCC regimens

6. Secondary Outcome: Disease Control Rate (DCR) Based on the Investigator's Radiographic Assessment
Description: DCR was defined as the percentage of patients who had a best overall response of CR, PR or at least 6 months with stable disease (SD). CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) with reduction in short axis to <10mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters while on study drug.
Time Frame: Date of randomization until data cutoff date of 21 August 2019 (up to 40 months)
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 67 | 66
Percentage of Participants | 13.4 [6.3 to 24.0] | 22.7 [13.3 to 34.7]
Statistical Analysis 1: Comparison: AGS-16C3F vs Axitinib; Test type: Superiority — A CMH analysis of the DCR, stratified for baseline ECOG-PS and number of prior systemic therapies for RCC, was conducted at a two-sided significance level of 0.05; p = 0.152, Cochran-Mantel-Haenszel — The stratified Mantel-Haenszel estimate of the odds ratio for experiencing objective response, with the axitinib arm as the reference level, was reported as a measure of relative treatment effect, along with its two-sided 95% CI; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.2 to 1.3]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: AE was defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures and which did not necessarily have a causal relationship with this treatment. An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, ECG data, and physical exam) was defined as an AE only if the abnormality induces clinical signs or symptoms or requires active intervention or requires interruption or discontinuation of study medication or the abnormality or investigational value is clinically significant in the opinion of the investigator. AE was considered "serious" if it results in death or is life threatening results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions or results in congenital anomaly, or birth defect requires inpatient hospitalization or leads to prolongation of hospitalization or other medically important events.
Time Frame: From first dose up to 53 months
Population: Safety Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | AGS-16C3F | Axitinib
Number analyzed (Participants) | 66 | 65
Participants | 65 | 64

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Antibody Drug Conjugate (ADC)
Description: Cmax of ADC was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: Pharmacokinetic Population (PKAS): (included all participants who were randomized to receive AGS-16C3F and had sufficient serum concentration data to facilitate derivation of at least 1 pharmacokinetic parameter, and for whom the time of dosing on the day of sampling was known) with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Microgram per Milliliter (μg/mL)
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 59
Microgram per Milliliter (μg/mL)
  Cycle 1 | 52.21 (58.407)
  Cycle 4: number analyzed (Participants) | 23
  Cycle 4 | 48.66 (38.820)

9. Secondary Outcome: Mean Predose Serum Concentration (Ctrough) of ADC
Description: Ctrough of ADC was reported.
Time Frame: Predose on cycle 2, 3, 4, 6, 14, and 18 (each cycle is 21 days)
Population: PKAS Population. Here, number of participants analyzed signifies participants who had quantifiable data.
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 50
Nanogram per Milliliter (ng/mL)
  Cycle 2 | 3429.39 (1402.334)
  Cycle 3: number analyzed (Participants) | 40
  Cycle 3 | 5194.21 (3602.012)
  Cycle 4: number analyzed (Participants) | 21
  Cycle 4 | 7731.38 (11171.906)
  Cycle 6: number analyzed (Participants) | 20
  Cycle 6 | 5695.13 (3899.222)
  Cycle 14: number analyzed (Participants) | 5
  Cycle 14 | 8698.26 (4239.327)
  Cycle 18: number analyzed (Participants) | 5
  Cycle 18 | 7213.32 (2082.501)

10. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of ADC
Description: Tmax of ADC was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 59
Days
  Cycle 1 | 0.04 [0.0 to 1.0]
  Cycle 4: number analyzed (Participants) | 23
  Cycle 4 | 0.05 [0.0 to 3.9]

11. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to 21days (AUC0 to 21) of ADC
Description: AUC (0 to 21) of ADC was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Day*Microgram per Milliliter (day*μg/mL)
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 52
Day*Microgram per Milliliter (day*μg/mL)
  Cycle 1 | 199.80 (68.821)
  Cycle 4: number analyzed (Participants) | 18
  Cycle 4 | 293.90 (100.190)

12. Secondary Outcome: Terminal Elimination Half-life (t1/2) of ADC
Description: t1/2 of ADC was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 49
Days
  Cycle 1 | 6.93 [3.9 to 19.6]
  Cycle 4: number analyzed (Participants) | 18
  Cycle 4 | 7.40 [3.6 to 14.5]

13. Secondary Outcome: Maximum Serum Concentration (Cmax) of Total Antibody (TAb)
Description: Cmax of TAb was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 59
μg/mL
  Cycle 1 | 37.49 (12.515)
  Cycle 4: number analyzed (Participants) | 23
  Cycle 4 | 42.84 (12.345)

14. Secondary Outcome: Mean Predose Serum Concnetration (Ctrough) of TAb
Description: Ctrough of TAb was reported.
Time Frame: Predose on cycle 2, 3, 4, 6, 14, and 18 (each cycle is 21 days)
Population: PKAS Population. Here, number of participants analyzed signifies participants who had quantifiable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 50
ng/mL
  Cycle 2 | 4966.69 (2571.410)
  Cycle 3: number analyzed (Participants) | 39
  Cycle 3 | 6943.11 (3666.956)
  Cycle 4: number analyzed (Participants) | 21
  Cycle 4 | 8660.94 (4176.472)
  Cycle 6: number analyzed (Participants) | 19
  Cycle 6 | 8777.51 (4131.388)
  Cycle 14: number analyzed (Participants) | 5
  Cycle 14 | 12491.90 (6593.131)
  Cycle 18: number analyzed (Participants) | 6
  Cycle 18 | 11726.15 (5572.172)

15. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of Tab
Description: Tmax of TAb was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 60
Days
  Cycle 1 | 0.05 [0.0 to 2.2]
  Cycle 4: number analyzed (Participants) | 23
  Cycle 4 | 0.05 [0.0 to 3.9]

16. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to 21days (AUC0 to 21) of TAb
Description: AUC (0 to 21) of TAb was reporetd.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 48
day*μg/mL
  Cycle 1 | 246.06 (88.815)
  Cycle 4: number analyzed (Participants) | 13
  Cycle 4 | 346.07 (158.029)

17. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Tab
Description: t1/2 of TAb was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 45
Days
  Cycle 1 | 8.70 [4.3 to 16.6]
  Cycle 4: number analyzed (Participants) | 13
  Cycle 4 | 9.15 [1.8 to 38.1]

18. Secondary Outcome: Maximum Serum Concentration (Cmax) of Cysteine Adduct of Maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF)
Description: Cmax of Cys-mcMMAF was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 64
ng/mL
  Cycle 1 | 6.09 (4.08)
  Cycle 4: number analyzed (Participants) | 25
  Cycle 4 | 3.78 (1.70)

19. Secondary Outcome: Mean Predose Serum Concnetration (Ctrough) of Cys-mcMMAF
Description: Ctrough of Cys-mcMMAF was reported.
Time Frame: Predose on cycle 2, 3, 4, 6, 14, and 18 (each cycle is 21 days)
Population: PKAS Population. Here, number of participants analyzed signifies participants who had quantifiable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 1
ng/mL
  Cycle 2: number analyzed (Participants) | 0
  Cycle 3: number analyzed (Participants) | 0
  Cycle 4: number analyzed (Participants) | 0
  Cycle 6 | 0.307 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Cycle 14: number analyzed (Participants) | 0
  Cycle 18: number analyzed (Participants) | 0

20. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of Cys-mcMMAF
Description: Tmax of Cys-mcMMAF was reported.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 64
Days
  Cycle 1 | 0.207 [0.139 to 0.954]
  Cycle 4: number analyzed (Participants) | 25
  Cycle 4 | 0.208 [0.197 to 1.11]

21. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to 21days (AUC0 to 21) of Cys-mcMMAF
Description: AUC (0 to 21) of Cys-mcMMAF was reporetd.
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point. Not calculated at cycle 4 due to an insufficient number of participants.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 21
day*ng/mL
  Cycle 1 | 9.61 (10.3)
  Cycle 4: number analyzed (Participants) | 0

22. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Cys-mcMMAF
Description: t1/2 of Cys-mcMMAF was reported
Time Frame: Predose, end of infusion, 4, 24, 72, 336 hours postdose of cycle 1 and cycle 4 (each cycle is 21 days)
Population: PKAS Population with available data at specified time point. Not calculated at cycle 4 due to an insufficient number of samples.
Measure: Median (Full Range); unit: Days
Arm/Group | AGS-16C3F
Number analyzed (Participants) | 1
Days
  Cycle 1 | 2.72 [2.72 to 2.72]
  Cycle 4: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose up to 53 months
Description: All-cause mortality data was reported for FAS population. Serious and non-serious adverse events were reported for safety population.
Arm/Group | AGS-16C3F | Axitinib
All-Cause Mortality (participants affected / at risk) | 36/67 | 44/66
Serious Adverse Events (participants affected / at risk) | 26/66 | 31/65
Other Adverse Events (participants affected / at risk) | 65/66 | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGS-16C3F (N=66) | Axitinib (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Device failure (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Craniotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGS-16C3F (N=66) | Axitinib (N=65)
Anaemia (Blood and lymphatic system disorders) | 15 (35) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (9) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 7 (8)
Diplopia (Eye disorders) | 4 (4) | 0 (0)
Dry eye (Eye disorders) | 14 (18) | 6 (6)
Eye pain (Eye disorders) | 7 (7) | 0 (0)
Photophobia (Eye disorders) | 5 (5) | 0 (0)
Vision blurred (Eye disorders) | 26 (38) | 7 (8)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 12 (20) | 10 (12)
Constipation (Gastrointestinal disorders) | 16 (16) | 21 (25)
Diarrhoea (Gastrointestinal disorders) | 12 (18) | 31 (70)
Dry mouth (Gastrointestinal disorders) | 6 (8) | 6 (10)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 7 (10)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 7 (8)
Nausea (Gastrointestinal disorders) | 31 (56) | 26 (40)
Oral pain (Gastrointestinal disorders) | 0 (0) | 5 (8)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 15 (23)
Vomiting (Gastrointestinal disorders) | 18 (25) | 22 (38)
Asthenia (General disorders) | 7 (8) | 5 (7)
Chills (General disorders) | 15 (29) | 2 (4)
Fatigue (General disorders) | 36 (48) | 37 (67)
Influenza like illness (General disorders) | 2 (2) | 5 (5)
Mucosal inflammation (General disorders) | 1 (1) | 5 (9)
Non-cardiac chest pain (General disorders) | 3 (3) | 4 (4)
Oedema peripheral (General disorders) | 11 (13) | 7 (10)
Pain (General disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 9 (18) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (7) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (16) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 5 (8) | 5 (7)
Blood bilirubin increased (Investigations) | 4 (10) | 2 (3)
Blood creatinine increased (Investigations) | 5 (8) | 5 (10)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 5 (5)
Platelet count decreased (Investigations) | 5 (9) | 2 (2)
Weight decreased (Investigations) | 7 (13) | 19 (30)
Decreased appetite (Metabolism and nutrition disorders) | 14 (17) | 24 (45)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 11 (15)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (6) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (23) | 24 (27)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 11 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 14 (22)
Dizziness (Nervous system disorders) | 14 (18) | 12 (16)
Dysgeusia (Nervous system disorders) | 3 (3) | 10 (11)
Headache (Nervous system disorders) | 16 (20) | 16 (23)
Memory impairment (Nervous system disorders) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 2 (2)
Tremor (Nervous system disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (6) | 5 (7)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Proteinuria (Renal and urinary disorders) | 1 (1) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 15 (20)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 25 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 18 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (23) | 5 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 7 (10)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (38)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (5)
Hypertension (Vascular disorders) | 4 (10) | 27 (48)
Hypotension (Vascular disorders) | 4 (6) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT02639182/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02639182/SAP_000.pdf